CLINICAL TRIAL: NCT02377011
Title: Randomised Controlled Trial of the Clinical and Cost Effectiveness of NICE Recommended Problem Solving Cognitive Behaviour Therapy (PS CBT) Delivered Remotely Versus Treatment as Usual in Adolescents and Young Adults With Depression Who Repeatedly Self-harm
Brief Title: RCT of the Clinical and Cost Effectiveness of Cognitive Behaviour Therapy (CBT) Delivered Remotely Versus Treatment as Usual in Adolescents and Young Adults With Depression Who Repeatedly Self-harm
Acronym: eDASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLAHRC-EM 14059
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2016-06

CONDITIONS: Depression and Self-Harm
MeSH Terms: conditions — Depression; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PS CBT (Experimental): Problem solving cognitive behaviour therapy (PS CBT) will be delivered remotely by means of telephone or video calling by a cognitive behaviour therapist in addition to their usual care.
  The duration of the intervention will be 10 sessions. Research measures will be completed at baseline, 3,6,9 and 12 months
  Interventions: Behavioral: Problem solving cognitive behaviour therapy (PS CBT)
- Treatment as Usual (No Intervention): Participants will not receive any CBT therapy in addition to their usual care. Research measures will be completed at baseline,3,6,9 and 12 months.

INTERVENTIONS:
Behavioral: Problem solving cognitive behaviour therapy (PS CBT)
  Arms: PS CBT

SUMMARY:
A randomized controlled trial to test the whether remote delivery of cognitive based therapy (CBT) is clinically and cost effective when compared to treatment as usual in adolescents and young adults with depression who self-harm.

DETAILED DESCRIPTION:
Self harm is one of the five leading causes of admission to acute hospital with rates increasing by nearly 50% from 2003-2009 (South West Public Health Observatory, 2012). Re-admission within 30 days is frequent. People who repeatedly self harm are at high risk for suicide and and as a result suicide, self-harm and crisis are priorities for CCGs and HWBs in the East Midlands.

The NICE Clinical Guideline 133 on longer-term treatment of self-harm recommends between 3 to 12 sessions of psychological treatment involving problem solving and alternative coping. Presently however, the biggest at risk group for self-harm and suicide is not offered any psychological treatment.

Studies have shown that mobile phones are a highly acceptable method of engaging adolescents with depression in psychological treatments such as CBT (Whittaker et al 2012). Furthermore a systematic review has show that treatment delivery via remote technology is just as effective as face-to-face in people with anxiety or depression (Bee et al, 2008).

The study therefore has the following aims and objectives:

1. To optimise and determine the acceptability and feasibility of engaging and retaining patients with depression who repeatedly self-harm in a remotely delivered (through video calling/telephone) CBT intervention over 10 sessions.
2. To outline the barriers and drivers to delivering both the study and the remotely delivered PS CBT intervention and how barriers to the interventions are addressed through a network of practice or other means.
3. If the recruitment and retention into the study and the remotely delivered PS therapy are feasible and acceptable, then we will determine the clinical effectiveness and cost effectiveness of the intervention versus treatment as usual.
4. If the intervention (pilot study) proves to be clinically effective and cost effective then the barriers and drivers to implementation in all counties in the East Midlands will be explored using a network of practice linking with NHS organisations, strategic clinical networks, and the AHSN (see qualitative analysis of barriers and drivers to the implementation of the intervention below).

The main hypothesis of this study is:

Adolescents and young adults who receive problem solving cognitive behaviour therapy (plus treatment as usual) will report greater reduction in their depressive symptoms (as measured using Beck depression inventory 2) from baseline to 6 months in comparison to those receiving treatment as usual.

Secondary objectives will be to observe a change over 12 months on measures of depression, hopelessness and suicidality.

Study configuration:

This study will compare two groups: participants will be randomly assigned to the TAU group (control group) or the remotely delivered PS CBT (and TAU) group (intervention group).

ELIGIBILITY:
Inclusion Criteria:

* >2 self-harm episodes.
* With high levels of unipolar depressive symptoms (BDI-2 score of 17 or more).
* Sufficient understanding of English (spoken and written).
* Ability to give informed consent

Exclusion Criteria:

* Clinical judgement of high level of suicide risk, other risk to self or others requiring other urgent approaches e.g. admission to mental health unit.
* Other severe mental illness e.g. psychosis, bipolar disorder, substance use disorder or organic mental disorder e.g. secondary to head injury as the primary mental health problem as determined by a structured psychiatric interview (SCID).
* Currently receiving structured psychological therapy

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (V2) | Baseline to 6 months
  The difference of change in self-rated depression as measured by Beck depression inventory (version 2) from baseline to 6 months, between the control and intervention group.

SECONDARY OUTCOMES:
Beck Depression Inventory (V2) | Baseline to 12 months
Time to Self-Harm | Baseline to 12 months
  Time to self-harm, assessed through a self-report measure and verified through medical records where possible
Patient Health Questionnaire 9 | Baseline to 12 months
  Depressive symptoms on the PHQ-9 (Kroenke et al, 2001)
Beck hopelessness scale | Baseline to 12 months
  Hopelessness measured on the Beck hopelessness scale (Beck, 1988)
Columbia Suicide Severity Rating Scale | Baseline to 12 months
  Suicidality measured on the Columbia Suicide Severity Rating Scale (CSSRS; Posner et al, 2011).
Social functioning | Baseline to 12 months
  Social functioning measured using the work and social adjustment scale (WSAS; Mundt et al, 2002).
Quality of life | Baseline to 12 months
  Quality of life measured using EQ-5D (EuroQol Group, 1990).
Cost Effectiveness | Baseline to 12 months
  A modified version of the Client Service Receipt Inventory (CSRI; Beecham & Knapp, 2001): to measure costs, service utilisation, income and related matters to analyse cost effectiveness.
Qualitative Interviews | Baseline to 12 months
  Explore reasons why individuals may or may not engage with the study and the PS CBT intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kapil Sayal, PhD, Principal Investigator — CLAHRC-EM, University of Nottingham
Locations (4):
- United Kingdom (4):
  - Derbyshire Healthcare NHS Foundation Trust, Derby, Derbyshire
  - Derbyshire Hoispitals NHS Foundation Trust, Derby, Derbyshire
  - Chesterfield Royal Hospital NHS Foundation Trust, Chesterfield, Deryshire
  - Nottinghamshire Healthcare NHS foundation Trust., Nottingham, Nottinghamshire

REFERENCES:
- [Background] Beck AT. Beck Hopelessness Scale. The Psychological Corporation: San Antonio, Texas, 1988.
- [Background] Beck AT, Steer RA, Brown GK. Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation, 1996.
- [Background] Bee PE, Bower P, Lovell K, Gilbody S, Richards D, Gask L, Roach P. Psychotherapy mediated by remote communication technologies: a meta-analytic review. BMC Psychiatry. 2008 Jul 22;8:60. doi: 10.1186/1471-244X-8-60. PMID 18647396
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Whittaker R, Merry S, Stasiak K, McDowell H, Doherty I, Shepherd M, Dorey E, Parag V, Ameratunga S, Rodgers A. MEMO--a mobile phone depression prevention intervention for adolescents: development process and postprogram findings on acceptability from a randomized controlled trial. J Med Internet Res. 2012 Jan 24;14(1):e13. doi: 10.2196/jmir.1857. PMID 22278284
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Sayal K, Roe J, Ball H, Atha C, Kaylor-Hughes C, Guo B, Townsend E, Morriss R. Feasibility of a randomised controlled trial of remotely delivered problem-solving cognitive behaviour therapy versus usual care for young people with depression and repeat self-harm: lessons learnt (e-DASH). BMC Psychiatry. 2019 Jan 24;19(1):42. doi: 10.1186/s12888-018-2005-3. PMID 30678674